CLINICAL TRIAL: NCT01871415
Title: A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PHASE III STUDY TO ASSESS THE EFFICACY, SAFETY AND TOLERABILITY OF ALEGLITAZAR PLUS METFORMIN COMBINATION THERAPY COMPARED WITH PLACEBO PLUS METFORMIN IN PATIENTS WITH TYPE 2 DIABETES MELLITUS INADEQUATELY CONTROLLED WITH METFORMIN MONOTHERAPY
Brief Title: A Study of Aleglitazar in Combination With Metformin in Patients With Type 2 Diabetes Mellitus Who Are Inadequately Controlled With Metformin Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YC28036
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aleglitazar + metformin (Experimental)
  Interventions: Drug: aleglitazar; Drug: metformin
- Placebo + metformin (Active Comparator)
  Interventions: Drug: metformin; Drug: placebo

INTERVENTIONS:
Drug: aleglitazar — 150 mcg orally daily
  Arms: Aleglitazar + metformin
Drug: metformin — pre-existing background regimen and dose
Drug: placebo — matching aleglitazar placebo orally daily
  Arms: Placebo + metformin

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the efficacy, safety and tolerability of aleglitazar in combination with metformin in patients with Type 2 diabetes mellitus who are inadequately controlled with metformin monotherapy. Patients will be randomized to receive either aleglitazar 150 mcg orally daily or placebo for 26 weeks in combination with their pre-existing metformin regimen and dose.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, >/= 18 years of age
* Type 2 diabetes mellitus treated with stable metformin monotherapy for at least 12 weeks prior to screening; metformin dose should be >/= 1500 mg/day (or individual maximum tolerated dose), but no more than the maximum dose specified in the label
* HbA1c >/= 7% and </= 9.5% at screening or within 4 weeks prior to screening and at pre-randomization visit
* Fasting plasma glucose </= 13.3 mmol/L (</= 240 mg/dL) at pre-randomization visit
* Agreement to maintain diet and exercise habits implemented during the run-in phase during the full course of the study

Exclusion Criteria:

* Pregnant women, women intending to become pregnant during the study period, currently lactating women, or women of child-bearing potential not using highly effective, medically approved birth control methods
* Diagnosis or history of:

  1. Type 1 diabetes mellitus, diabetes resulting from pancreatic injury, or secondary forms of diabetes
  2. Acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma within the past 6 months
* Any previous treatment with thiazolidinedione or with a dual PPAR agonist
* Any body weight lowering or lipoprotein-modifying therapy (e.g. fibrates) within 12 weeks prior to screening with the exception of stable (>= 1 month) statin therapy
* Prior intolerance to fibrate
* Treatment with anti-diabetic medication other than metformin in the last 12 weeks prior to screening
* Triglycerides (fasting) > 4.5 mmol/L (> 400 mg/dL) at screening or within 4 weeks prior to screening
* Clinically apparent liver disease
* Anemia at or within 4 weeks prior to screening
* Inadequate renal function
* Symptomatic congestive heart failure NYHA Class II-IV at screening
* Myocardial infarction, acute coronary syndrome or transient ischemic attack/stroke within 6 months prior to screening visit
* Known macular edema at screening or prior to screening visit
* Diagnosed and/or treated malignancy (except for basal cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) within the past 5 years
* Uncontrolled hypertension
* History of active substance abuse (including alcohol) within the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to Week 26

SECONDARY OUTCOMES:
Change in lipids | from baseline to Week 26
Change in fasting plasma glucose (FPG) | from baseline to Week 26
Responder rates, defined as target HbA1c: < 7.0%, < 6.5% at Week 26 | 26 weeks
Change in homeostatic index of insulin sensitivity (by HOMA-IS) | from baseline to Week 26
Change in homeostatic index of beta cell function (by HOMA-BFC) | from baseline to Week 26
Change in markers of insulin sensitivity/cardiovascular risk | from baseline to Week 26
Safety: Incidence of adverse events | approximately 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- China (4):
  - Shanghai
  - Shenyang
  - Shiyan
  - Suzhou
- South Korea (3):
  - Gyeonggi-do
  - Incheon
  - Seoul